CLINICAL TRIAL: NCT01747226
Title: Masking and Therapeutic Effect of Different Mouth Rinses in Patients With Oral Malodor.
Brief Title: Effect of Mouth Rinses in Oral Malodor
Acronym: MR2012
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Gaba International AG (Industry)
Responsible Party: Principal Investigator, Marc Quirynen, PhD DDS, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GASAS-1205X
Record Dates: First submitted 2012-12-05; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Halitosis
Keywords: Oral malodor; Halitosis; Bad Breath; Mouth rinses; Mouthwashes; Amine fluoride/Stannous fluoride; Zinc ions; Chlorhexidine
MeSH Terms: conditions — Halitosis | interventions — Water; Drinking Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fluoride rinse (Placebo Comparator): A fluoride rinse with alcohol was chosen because its similarity in color and aroma to the active rinses. This anti-cavity rinse does not contain any active components and therefore it is not expected to have any anti-malodour activity.
  Interventions: Other: Fluoride rinse
- Halita (Active Comparator): Halita is a CHX-containing benchmark product that has proven to be clinically effective against halitosis (Roldan et al, 2003)
  Interventions: Other: Halita
- Meridol Halitosis (Active Comparator): This study aims to confirm the effect of meridol®Halitosis(AmF/SnF2 and zinc) already observed in volunteers with morning bad breath (physiological)(Wigger-Alberti et al, 2010; Wilhelm et al, 2010)in patients with oral malodor (pathological).
  Interventions: Other: Meridol Halitosis
- Water (Sham Comparator): To distinguish the masking effect caused by the formulations and the one caused by the rinsing itself.Only for short term evaluation (15') to not to compromise compliance of patients.
  Interventions: Other: Water

INTERVENTIONS:
Other: Fluoride rinse — rinse with 15 ml for 1 minute
  Arms: Fluoride rinse
Other: Halita — rinsing with 15 ml for 1 minute
  Other Names: - Halita mouthwash 500 ml. CN 323923.3; - Halita, Dentaid Spain
  Arms: Halita
Other: Meridol Halitosis — rinsing with 15 ml for 1 minute
  Other Names: name of product meridol® HALITOSIS mouthrinse; GABA product number:266831; PDM number: 3*21750; name of manufacturer:GABA International AG
  Arms: Meridol Halitosis
Other: Water — rinsing with 15ml for 1 minute
  Other Names: bottled water
  Arms: Water

SUMMARY:
Bad breath or halitosis is caused by specific gases originating from the mouth or the expired air. In most cases the pathology lies within the mouth and in this case receives the name pathologic halitosis of oral cause or oral malodor. The aim of this study is to evaluate the immediate (masking) and long term (therapeutic) effect of commercially available mouth rinses in the treatment of oral malodor. For this volunteers with oral malodor detected by organoleptic evaluation and confirmed by the increase level of sulphur compounds in their breath (VSC) will be asked to use a designated mouthwash. The breath parameters will be assessed at baseline and 15' after the first rinse (15 ml, during 1 minute) and over night at the end of a period of 3 weeks during which the volunteers rinsed twice a day (15 ml, 1 minute) with the assigned mouthwash. The short and long term effect of a stannous fluoride/amine fluoride/zinc rinse; a chlorhexidine/cetylpyridinium chloride/zinc product and a negative control(fluoride rinse and/or water) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Age ≥ 18 years
* Organoleptic score of breath ≥ 2
* VSC readings (sum of H2S and CH3SH by OralChroma) ≥ 120 ppb*
* Intra-oral cause of bad breath
* Non-smokers
* Willing to participate and able to give written informed consent

Exclusion Criteria:

* Ongoing dental treatment or any other medical treatment of the oral cavity
* Any known allergy to previously used oral hygiene products or any known allergy to any of the ingredients of the study products, which are used during the study
* Any pathological change of the oral mucosa
* Use of prohibited treatments / therapies and/or abuse of drugs, alcohol, etc
* Pregnancy or breastfeeding
* Active caries
* Acute sinusitis
* Severe oro-pharyngeal infections
* On medications which can cause malodour
* Reduced salivary flow due to pathological reasons (e.g. Sjögren syndrome)
* Situation considered not compatible with the study according to the investigator's opinion; the latter includes: patients eating very spicy food, persons under homeopathic therapy, patients who used antibiotics during the 2 months before the study, patients frequently using chewing gum, patients under corticosteroids or other serious medications.
* Patients unwilling to abstain from additional oral hygiene (only toothbrushing allowed) particularly mouthrinse, chewing gums, breath strips, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline organoleptic score of breath (OLS) | after15' and after 3 weeks
  A trained and calibrated "judge" sniffs the expired air of the volunteer and assesses whether it is unpleasant by using an intensity rating, normally from 0 to 5, with 0 = no odor present, 1 = barely noticeable odor, 2 = slight but clearly noticeable odor, 3 = moderate odor, 4 = strong offensive odor, and 5 = extremely foul odor (proposed by Rosenberg and McCulloch.
Change from baseline in H2S and CH3SH level in breath | after 15' and after 3 weeks
  A portable gas chromatograph (OralChroma™, Abilit Corporation, Kanagawa, Japan) will be used to measures the concentration of hydrogen sulphur (H2S) and methyl mercaptan (CH3SH) in mouth air. The device has been calibrated and validated for its use by the manufacturer.

SECONDARY OUTCOMES:
Change from baseline global level of volatile sulphur compounds (VSC) | after 15' and after 3 weeks
  A portable device (Halimeter®, Interscan Corporation, model RH-17E, Chatsworth, USA)able to detect sulphur compounds in air will be used according to the manufacturer instructions
Change from baseline microbial load of saliva | after 3 weeks
  A sample of non-stimulated saliva will be collected into a sterile container and kept at 4°C till processing. To the standard culture of the samples (of aerobic and anaerobic incubation at 37°C) a molecular technique (qPCR)of bacterial detection will be added for periodontal pathogens (P. gingivalis, P intermedia, F. nucleatum and A. actinomycetemcomitans) and bacteria usually involved in oral malodour (S. moorei).
Change from baseline microbial load of tongue coating | after 3 weeks
  Tongue coating will be collected by wiping a sterile swab 3 times over the dorsum of the tongue, in the area of the foramen caecum. Till analysis; the tip of the cotton swab will be kept in a vial containing 2ml of reduced transport fluid (RTF). To the standard culture of the samples (of aerobic and anaerobic incubation at 37°C) a molecular technique (qPCR)of bacterial detection will be added for periodontal pathogens (P. gingivalis, P intermedia, F. nucleatum and A. actinomycetemcomitans) and bacteria usually involved in oral malodour (S. moorei).

OTHER OUTCOMES:
Patients' opinion | after 3 weeks
  Patients' opinion regarding product satisfaction will be scored on a VAS line (0 to 10). The questionnaire will include the following points:satisfaction, side effects, use, future use and effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Quirynen, PhD, DDS, Principal Investigator — Universitarie Ziekenhuis Leuven
Locations (1):
- Department of Periodontology, KULeuven, Leuven, Belgium

REFERENCES:
- [Background] Quirynen M, Dadamio J, Van den Velde S, De Smit M, Dekeyser C, Van Tornout M, Vandekerckhove B. Characteristics of 2000 patients who visited a halitosis clinic. J Clin Periodontol. 2009 Nov;36(11):970-5. doi: 10.1111/j.1600-051X.2009.01478.x. Epub 2009 Oct 6. PMID 19811581
- [Background] Wilhelm D, Gysen K, Himmelmann A, Krause C, Wilhelm KP. Short-term effect of a new mouthrinse formulation on oral malodour after single use in vivo: a comparative, randomized, single-blind, parallel-group clinical study. J Breath Res. 2010 Sep;4(3):036002. doi: 10.1088/1752-7155/4/3/036002. Epub 2010 Aug 17. PMID 21383479
- [Background] Wigger-Alberti W, Gysen K, Axmann EM, Wilhelm KP. Efficacy of a new mouthrinse formulation on the reduction of oral malodour in vivo. A randomized, double-blind, placebo-controlled, 3 week clinical study. J Breath Res. 2010 Mar;4(1):017102. doi: 10.1088/1752-7155/4/1/017102. Epub 2009 Dec 18. PMID 21386207